CLINICAL TRIAL: NCT04042896
Title: Effects of Exergame vs. Traditional Aerobic Exercise in Patients at High Cardiovascular Risk
Brief Title: Effects of Exergame in Patients at High Cardiovascular Risk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoung Im Cho (Other)
Responsible Party: Sponsor-Investigator, Kyoung Im Cho, Clinical Professor, Kosin University Gospel Hospital
Organization: Kosin University Gospel Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EXERHEART
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Aerobic Exercise; Cardiorespiratory Fitness; Cardiovascular Diseases
Keywords: Aerobic exercise; Exergame; cardiorespiratory fitness; endothelial function; epicardial fat
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: exergame group, treadmill group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exergame group (Experimental): The exergame group performed exercise using the Exer Heart device (D&J Humancare, Seoul, South Korea), which consisted of a running/jumping board and a screen connected to the board. The exercise program "Alchemist's Treasure", a running-based exergame, moves the avatar according to the user's motions and was used for the exercise session. "Alchemist's Treasure" is a game in which the user listens to stimulating music, runs with the avatar, avoiding obstacles, and wins items using the front, back, left, and right sensors on the exercise board. The subject can control the speed of the avatar movement by adjusting the walking or running speed on the board.
  This study did not enforce exercise intensity in order to allow patients to enjoy the exergame. Thus, during the training period, the patients exercised at a self-selected pace for 40 minutes per day.
  Interventions: Behavioral: exergame
- treadmill group (Active Comparator): The treadmill group consisted of 40 minutes of walking or jogging at 60-80% of the heart rate (HR) reserve. The exercise intensity was determined using the Karvonen method target HR = [Exercise Intensity × (HRmax - resting HR)] + resting HR. The HR was recorded during each session using an HR monitor (Polar RS400sd; Madison Height, Michigan, USA). The control group was asked to maintain their regular physical activity level for 12 weeks.
  Interventions: Behavioral: treadmill exercise
- control group (No Intervention): The control group was asked to maintain their regular physical activity level for 12 weeks.

INTERVENTIONS:
Behavioral: exergame — Exergame is 'exercise + game'.
  Arms: exergame group
Behavioral: treadmill exercise — traditional aerobic exercise
  Arms: treadmill group

SUMMARY:
Background: Exergaming is thought to have a similar effect on cardiovascular (CV) responses as aerobic fitness activities. The aim of this study was to compare the cardiovascular effects of exergaming and traditional treadmill exercises in patients with high CV risk.

Methods: Sixty-four patients with high CV risk were randomized among exergame (EG: n = 22), treadmill (TM: n = 22), and control (n=20) groups. The EG group was engaged in the running-based exergame using Exer Heart and the TM group walked or jogged on a treadmill. Cardiorespiratory fitness (CRF), brachial artery flow-mediated dilation (FMD), endothelial progenitor cell numbers (EPCs), epicardial fat thickness (EFT), metabolic parameters and anthropometric parameters were measured in patients before and 3 months after the training.

DETAILED DESCRIPTION:
Introduction Cardiovascular (CV) disease is a major cause of premature death and morbidity worldwide. It is widely known that age, sex, hypertension, dyslipidemia, diabetes, and smoking are the main risk factors which can cause CV disease[1]. Many other CV risk factors and their markers have been identified in recent studies. Among these, cardiorespiratory fitness (CRF) and endothelial dysfunction are strong predictors of the risk of developing CV disease[2, 3]. In addition, epicardial adipose tissue is a visceral fat which accumulates in the epicardium of the heart, and has recently been considered as a new index of CV risk[4, 5].

It is well established that regular exercise (physical activity) is effective in preventing and treating CV risk factors by improving health-related fitness[6]. Despite the health benefits of regular exercise, many patients with CV risk factors often do not participate in regular exercise for reasons including lack of time, motivation, or interest.

In recent years, a new exercise program called exergame has been developed as a result of the technical advancements in gaming and virtual reality programs. Exergames are interactive video games which provide the opportunity to increase physical activity by requiring movement of the entire body[7] and are proving to be an alternative exercise modality. In addition, exergames are used to fight pediatric obesity[8], improve senior physical performance[9], and facilitate poststroke motor rehabilitation[10]. However, only a few studies have examined the effects of exergaming on CV or chronic disease related risk factors. Furthermore, in order for exergames to progress as a rehabilitation program for the prevention and treatment of CV disease in the future, it is necessary to compare it to traditional aerobic exercises.

Therefore, the aim of this study was to compare the effects of exergame versus treadmill exercises on cardiorespiratory fitness (CRF), endothelial function, epicardial fat, cardiometabolic, and anthropometric parameters in patients with high CV risk.

Methods Participants and Study Design This single-center study was approved by the Institutional Review Board of Kosin University Gospel Hospital (Protocol no. KUGH 2016-06-029). Sixty-four female patients with a Framingham CV disease 10-year risk score above 20% were enrolled in this study[11, 12]. All participants voluntarily participated in the study and signed a consent form agreeing to the study process. In order to reduce the margin of error due to sex differences and physiological responses to the greatest degree possible, only post-menopausal women were recruited considering the hormonal changes which occur during menstruation. The inclusion criteria were post-menopausal women aged ≤80 years who did not have a history of participating in regular exercise within the past 3 months. The exclusion criteria were resistant hypertension, any systemic disease including significant liver disease, neurologic disorders, malignant disease, renal failure, chronic obstructive pulmonary disease, valvular heart disease, a positive treadmill test, a history of acute coronary syndrome, myocardial infarction or any revascularization procedure, or musculoskeletal patients for whom exercise was impossible. Patients were randomized to the exergame (EG: n=22), treadmill (TM: n=22), or control (n=20) groups.

All subjects were tested over a two-day period before and after 3 months of training. On the first visit, the subject's height, weight, waist circumference (WC), blood sampling, and blood pressure (BP) were obtained after 8 hours of fasting. On the second visit, brachial artery flow mediated dilatation (FMD), epicardial fat thickness (EFT) measured by echocardiography, and CRF tests were performed after 4 hours fasting. In addition, subjects were asked to refrain from excessive exercise, overeating, and caffeine consumption for 24 hours before all tests.

Cardiorespiratory Fitness CRF was assessed using a treadmill testing protocol[13]. The test was carried out on a programmable treadmill (GE CASE T2100; GE Medical Systems, Milwaukee, WI, USA) using a Ramp protocol until exhaustion in a temperature-controlled room (21-23°C). The cardiac rhythm was continuously monitored with a 12-lead electrocardiogram system. BP monitoring was carried out using an automated device (Suntech Tango; Suntech Medical, Morrisville, NC, USA). Ventilation (VE), oxygen uptake (VO2), and carbon dioxide output (VCO2) were measured using a computerized system (Cosmed K4b2, Cosmed Ltd., Rome, Italy). The termination of the test occurred when the subject's rated perceived exertion (RPE) was greater than 17, the respiratory exchange ratio was greater than 1.05, the oxygen intake had plateaued despite an increased workload, or the subject requested test termination. The highest recorded oxygen intake was defined as the VO2 peak of each person.

Flow-Mediated Dilation FMD was measured in the brachial artery according to current guidelines[14]. After the subject had relaxed sufficiently for 10 to 20 minutes in the supine position, the baseline value was measured. Two-dimensional ultrasonography (Vivid 7; General Electric, Horten, Norway) was performed using a 10-MHz linear-array transducer probe. After the baseline measurement, reactive hyperemia was induced by the inflation of a pneumatic cuff to 180-200 mmHg (50 mmHg higher than SBP) for five minutes on the forearm. For the peak diameter of the brachial artery, the diameter was recorded 40-60-seconds after sudden deflation of the cuff. The percent FMD induced by reactive hyperemia was expressed as the relative change from baseline (%FMD = 100 × [diameter after hyperemia-baseline diameter]/baseline diameter). At the peak of the R wave of the surface electrocardiogram, each diameter was measured three times during two heartbeats and the average values were used for the final analysis.

Epicardial Fat Thickness Epicardial adipose tissue was measured by assessing EFT through echocardiography[15]. Echocardiographic assessment of the EFT was defined as the echo-free space between the outer wall of the myocardium and the visceral layer of the pericardium. Standard 2-dimensional echocardiography was performed with the subject in the left lateral decubitus position using a 3.5 MHz transducer (Philips iE33, Philips Medical Systems, Bothell, WA, USA). The echocardiographic EFT test was conducted vertically from the free wall of the right ventricle at the end-systolic point in 3 heart cycles. One of the major problems with EFT measurements is the inconsistency of measurement locations. Therefore, in this study, the EFT value was recorded by considering the average of the parasternal long axis, parasternal short axis, and apical 4-chamber view. In addition, to minimize observational bias in a priori and post-hoc analyses, the researcher was blinded to the baseline value.

Exercise Training The EG group performed exercise using the Exer Heart device (D&J Humancare, Seoul, South Korea), which consisted of a running/jumping board and a screen connected to the board (Figure 1). The exercise program "Alchemist's Treasure", a running-based exergame, moves the avatar according to the user's motions and was used for the exercise session. "Alchemist's Treasure" is a game in which the user listens to stimulating music, runs with the avatar, avoiding obstacles, and wins items using the front, back, left, and right sensors on the exercise board (Figure 2). The subject can control the speed of the avatar movement by adjusting the walking or running speed on the board. Furthermore, the Exer Heart game does not harm the joints, as the activities are performed on the exercise board's soft material.

The exergame cannot continuously maintain intensity by fixing the speed and inclination like a treadmill motion due to the characteristics of the program. On the other hand, the biggest advantage of the exergame is enjoyment. This study did not enforce exercise intensity in order to allow patients to enjoy the exergame. Thus, during the training period, the patients exercised at a self-selected pace for 40 minutes per day. Instead, we monitored individual exercise intensity by monitoring HR (Polar RS400sd; Madison Height, Michigan, USA) and recorded the resting, minimum, maximum, and average HR during the exergame training period. The resting HR of the patients was 79 ± 12 beats per minute (bpm), the minimum HR was 98 ± 26 bpm, the maximum HR was 153 ± 28 bpm, and the mean HR was 120 ±19. According to the guidelines of the American College of Sports Medicine (ACSM), the range of exercise intensity for exergaming is between 42% and 82% of HR reserve.

The TM group consisted of 40 minutes of walking or jogging at 60-80% of the heart rate (HR) reserve. The exercise intensity was determined using the Karvonen method target HR = [Exercise Intensity × (HRmax - resting HR)] + resting HR. The HR was recorded during each session using an HR monitor (Polar RS400sd; Madison Height, Michigan, USA). The control group was asked to maintain their regular physical activity level for 12 weeks.

Exercise training was conducted at the Kosin University Gospel Hospital U-Healthcare Center. All subjects were engaged in exercise training under the expert supervision of a director and were trained to immediately notify the director of any abnormal symptoms during the exercise training and to consult a doctor if needed. For both the EG and TM groups, exercise training was comprised of a 5 minute warm-up, a 40 minute main exercise, and a 5 minute cool-down. After a necessary 2 week initial adjustment period, the exercise training was conducted 3 times per week for 12 weeks. Subjects who did not perform more than 80% of the 12 week exercise program were excluded from this study.

Statistical Analysis All values are presented as the mean ± standard deviation (SD). We used the chi-square test for category type variables. The paired t-test was used to compare the baseline and data after the 12 week exercise intervention for each group. One-way ANOVA with repeated measures (group × time) was used to compare the data between groups. Bonferroni post-hoc analysis was performed to evaluate the differences among groups. Pearson's correlation was used to evaluate the relationship between variables. Statistical significance was set to p<0.05. For statistical analysis, SPSS 21.0 (SPSS, Chicago, IL, USA), a statistical program for Windows, was used.

ELIGIBILITY:
Inclusion Criteria:

* Framingham CV disease 10-year risk score above 20%
* post-menopausal women
* no history of exercise

Exclusion Criteria:

* resistant hypertension
* liver disease
* neurologic disorders
* malignant disease
* chronic obstructive pulmonary disease
* valvular heart disease
* musculoskeletal patients

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change of volume of maximal oxygen uptake | Change from Baseline maximal oxygen uptake at 3 months
  maximal oxygen uptake refers to the ability of the circulatory and respiratory systems to supply oxygen to skeletal muscles during sustained physical activity.

SECONDARY OUTCOMES:
Change of percent of flow mediated dilation | Change from Baseline flow mediated dilation at 3 months
  Flow-mediated dilation (FMD) refers to dilation (widening) of an artery when blood flow increases in that artery. The primary cause of FMD is release of nitric oxide by endothelial cells.
  To determine FMD, brachial artery dilation following a transient period of forearm ischemia is measured using ultrasound. Because the value of FMD can be compromised when improperly applied, attempts have been made to standardize the methodology for measuring FMD.
Change of thickness of epicardial adipose tissue | Change from Baseline epicardial adipose tissue at 3 months
  Epicardial adipose tissue (EAT) is a particular form of visceral fat deposited around the heart and found to be a metabolically active organ that generates various bioactive molecules, which might significantly affect cardiac function. Marked component differences have been observed in comparing EAT with subcutaneous fat, suggesting a depot specific impact of stored fatty acids on adipocyte function and metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Im Cho, MD, PhD, Principal Investigator — Kosin University Gospel Hospital
Locations (1):
- Kosin University Gospel Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baranowski T, Abdelsamad D, Baranowski J, O'Connor TM, Thompson D, Barnett A, Cerin E, Chen TA. Impact of an active video game on healthy children's physical activity. Pediatrics. 2012 Mar;129(3):e636-42. doi: 10.1542/peds.2011-2050. Epub 2012 Feb 27. PMID 22371457